CLINICAL TRIAL: NCT06552832
Title: Clinician-Assisted Video Feedback Exposure-Approach Therapy (CAVEAT): An Open-Trial of a Brief Psychotherapy for Traumatized Mothers and Their Young Children
Brief Title: CAVEAT: An Open-Trial Feasibility Study
Acronym: CAVEAT-OT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Sandra Rusconi Serpa (Unknown)
Responsible Party: Principal Investigator, Daniel Schechter, Associate Professor and Senior Consultant in Child & Adolescent Psychiatry, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-SUPEA-01
Record Dates: First submitted 2024-05-06; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Parent-Child Relations; PTSD; Dissociation
Keywords: Brief Psychotherapy; Videofeedback; Mentalization; Infant Mental Health; Parenting; Interpersonal Violence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Dissociative Disorders

STUDY DESIGN:
Intervention Model Description: Open Trial with Pre- and Post-Measures (Treatment as Usual as parallel contrast without randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAVEAT (Experimental): Clinician-Assisted Videofeedback Exposure
  Interventions: Other: CAVEAT

INTERVENTIONS:
Other: CAVEAT — Brief manualized parent-child psychotherapy

SUMMARY:
This is an open-clinical trial to study the feasibility of a brief manualized psychotherapy for mothers interpersonal violence-related posttraumatic stress disorder (PTSD) and their very young children ages 1-3 years, entitled: Clinician-Assisted Videofeedback Exposure Approach Therapy (CAVEAT). This project, to be conducted with referred mothers and children to an academic medical center ambulatory care setting, intends to pilot along with the manualized intervention, pre- and post-intervention measures for up to 10 dyads over 2 years.

DETAILED DESCRIPTION:
This study is based on empirical research findings that demonstrate psychobiological dysregulation at multiple levels among violently traumatized mothers of infants and young children. A number of studies over the past decades have described the deleterious effects this dysregulation can have on the mother-infant relationship during formative development of self-regulation of emotion, arousal, and aggression in the young child. Out of this research and clinical experience, the principal investigator (PI) developed The Clinician-Assisted Videofeedback Exposure Session (CAVES) originally as an experimental evaluation technique and test-intervention (Schechter, 2003). The theoretical premise, evidence-base, and signature features of the CAVES became the foundation for a new brief psychotherapeutic model for traumatized parents and their very young children ages 1 to 4, Clinician-Assisted Videofeedback Exposure Approach Therapy (CAVEAT). Two published studies involving both a clinically-referred and non-referred sample of mothers and children have shown a significant reduction in the degree of negativity and age-inappropriateness of maternal attributions towards her child (Schechter et al., 2006; Schechter et al., 2015). The latter is important as maternal attributions represent "keys" to maternal mental representations that, in turn, mark the mother's transference to her own child (Lieberman, 1999). Lacking thus far, however, has been a study to examine the sustainability of these changes in maternal perception and whether change in maternal perception translates into measurable change in mother-child interactive behaviour including increased maternal sensitivity, reflective functioning, and reduction in child symptoms. Since 2008, the PI has closely collaborated on a number of projects with the co-PI, who has extensive experience in psychotherapy research having worked with pioneers Bertrand Cramer, Daniel Stern in Switzerland (Cramer et al., 1990) and Susan McDonough in the US (Rusconi Serpa, Sancho Rossignol, & McDonough, 2009). In 2012, the PI, co-PI and colleagues began to conceptualize a manualized brief-psychotherapy that would be most likely to sustain changes over time: CAVEAT. Sessions are divided into 4 modules: 1. Evaluation, diagnostic formulation, and identification of objectives and triggers of maternal posttraumatic stress in the parent-child relationship (5 sessions); 2. Differentiation between past and present relationships (4 sessions);

ELIGIBILITY:
Inclusion Criteria:

* French-speaking, biological child living with mother

Exclusion Criteria:

* Physical and/or mental handicap that can interfere with participation in play and measures, active psychotic illness or substance abuse

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index- Short Form | Pre- and Post-Intervention within 6 weeks after last session
  Self-report questionnaire
Maternal Attributions Rating Scale | Pre- and Post-Intervention within 6 weeks after last session
  Clinician-rated measure
Brief Infant-Toddler Social Emotional Assessment | Pre- and Post-Intervention within 6 weeks after last session
  Maternal-report questionnaire

SECONDARY OUTCOMES:
Intervention Satisfaction Questionnaire | Post-Intervention within 6 weeks after last session
  Maternal and Therapist completed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Child & Adolescent Psychiatry Service, Lausanne, Canton of Vaud, Switzerland